CLINICAL TRIAL: NCT01975220
Title: Relative Bioavailability of Two Newly Developed FDC Tablet Strengths (25mg/1000mg and 12.5mg/750mg) of Empagliflozin/Metformin Extended Release Compared With the Free Combination of Empagliflozin and Metformin Extended Release in Healthy Subjects (an Open-label, Randomised, Single Dose, Two-way Crossover Study)
Brief Title: Relative Bioavailability of 2 Fixed Dose Combinations of Empagliflozin/Metformin Compared With Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.13
Record Dates: First submitted 2013-10-29; First posted 2013-11-04 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2016-08

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

ARMS (3):
- High dose, fasted (Experimental): 1 fixed dose combination (FDC) tablet vs. 3 single tablets under fasted conditions
  Interventions: Drug: 25 mg Empagliflozin/1000 mg Metformin XR, FDC; Drug: 1 tablet Empagliflozin/2 tablets Metformin XR
- High dose, fed (Experimental): 1 fixed dose combination (FDC) tablet vs. 3 single tablets under fed conditions
  Interventions: Drug: Empagliflozin/Metformin XR, FDC; Drug: 1 tablet Empagliflozin/2 tablets Metformin XR
- Low dose, fasted (Experimental): 2 fixed low dose combination (FDC) tablets vs. 4 single tablets under fed conditions
  Interventions: Drug: Empagliflozin/Metformin XR FDC; Drug: 1 tablet Empagliflozin/3 tablets Metformin XR

INTERVENTIONS:
Drug: Empagliflozin/Metformin XR, FDC — Experimental: high dose empagliflozin/metformin XR, FDC tablet
  Arms: High dose, fed
Drug: Empagliflozin/Metformin XR FDC — Experimental: low dose empagliflozin/metformin XR, FDC tablet
  Arms: Low dose, fasted
Drug: 25 mg Empagliflozin/1000 mg Metformin XR, FDC — Experimental, high dose Empagliflozin/Metformin XR,FDC Tablet
  Arms: High dose, fasted
Drug: 1 tablet Empagliflozin/2 tablets Metformin XR — Active Comparator: 1x empagliflozin/2x metformin XR tablets
  Arms: High dose, fasted
Drug: 1 tablet Empagliflozin/3 tablets Metformin XR — Active Comparator: 1x empagliflozin/3x metformin XR tablets
  Arms: Low dose, fasted
Drug: 1 tablet Empagliflozin/2 tablets Metformin XR — Active Comparator: 1x empagliflozin/2x metformin XR tablets
  Arms: High dose, fed

SUMMARY:
The purpose of this trial is to demonstrate the relative bioavailability of 2 newly developed fixed dose combination (FDC) tablets containing empagliflozin & metformin and the single tablets of empagliflozin and metformin when administered singularly.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males or females
2. Age 18-50 years (incl)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl)
4. Subjects must be able to understand and comply with study requirements

Exclusion criteria:

Any deviation from healthy condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.13.1 Boehringer Ingelheim Investigational Site, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose, Fasted: 1 FDC Tablet First, Then 3 Single Tablets: 1 fixed dose combination (FDC) tablet first, then 3 single tablets under fasted conditions:
  25 mg Empagliflozin/1000 mg Metformin extended release (XR), FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet;
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets
- High Dose, Fasted: 3 Single Tablets First, Then 1 FDC Tablet: 3 single tablets first, then 1 fixed dose combination (FDC) tablet under fasted conditions:
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets;
  25 mg Empagliflozin/1000 mg Metformin XR, FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet
- High Dose, Fed: 1 FDC Tablet First, Then 3 Single Tablets: 1 fixed dose combination (FDC) tablet first, then 3 single tablets under fed conditions:
  25 mg Empagliflozin/1000 mg Metformin XR, FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet;
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets
- High Dose, Fed: 3 Single Tablets First, Then 1 FDC Tablet: 3 single tablets first, then 1 fixed dose combination (FDC) tablet under fed conditions:
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets;
  25 mg Empagliflozin/1000 mg Metformin XR, FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet
- Low Dose, Fasted: 2 FDC Tablets First, Then 4 Single Tablets: 2 fixed low dose combination (FDC) tablets first, then 4 single tablets under fasted conditions:
  12.5 mg Empagliflozin / 750 mg Metformin XR FDC tablets: Experimental: low dose Empagliflozin/Metformin XR, 2 FDC tablets;
  1 x 25 mg tablet Empagliflozin / 3 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 3x Metformin XR tablets
- Low Dose, Fasted: 4 Single Tablets First, Then 2 FDC Tablets: 4 single tablets first, then 2 fixed low dose combination (FDC) tablets under fasted conditions:
  1 x 25 mg tablet Empagliflozin / 3 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 3x Metformin XR tablets;
  12.5 mg Empagliflozin/750 mg Metformin XR FDC tablets: Experimental: low dose Empagliflozin/Metformin XR, 2 FDC tablets
Period: Test Period 1
Arm/Group | High Dose, Fasted: 1 FDC Tablet First, Then 3 Single Tablets | High Dose, Fasted: 3 Single Tablets First, Then 1 FDC Tablet | High Dose, Fed: 1 FDC Tablet First, Then 3 Single Tablets | High Dose, Fed: 3 Single Tablets First, Then 1 FDC Tablet | Low Dose, Fasted: 2 FDC Tablets First, Then 4 Single Tablets | Low Dose, Fasted: 4 Single Tablets First, Then 2 FDC Tablets
Started | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 11 | 12 | 12 | 12 | 12
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Not treated | 0 | 1 | 0 | 0 | 0 | 0
Period: Test Period 2
Arm/Group | High Dose, Fasted: 1 FDC Tablet First, Then 3 Single Tablets | High Dose, Fasted: 3 Single Tablets First, Then 1 FDC Tablet | High Dose, Fed: 1 FDC Tablet First, Then 3 Single Tablets | High Dose, Fed: 3 Single Tablets First, Then 1 FDC Tablet | Low Dose, Fasted: 2 FDC Tablets First, Then 4 Single Tablets | Low Dose, Fasted: 4 Single Tablets First, Then 2 FDC Tablets
Started | 12 | 11 | 12 | 12 | 12 | 12
Completed | 12 | 11 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug.
Groups:
- High Dose, Fasted: 1 fixed dose combination (FDC) tablet vs. 3 single tablets under fasted conditions:
  25 mg Empagliflozin/1000 mg Metformin XR (extended release), FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet;
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets
- High Dose, Fed: 1 fixed dose combination (FDC) tablet vs. 3 single tablets under fed conditions:
  25 mg Empagliflozin/1000 mg Metformin XR, FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet;
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets
- Low Dose, Fasted: 2 fixed low dose combination (FDC) tablets vs. 4 single tablets under fasted conditions:
  12.5 mg Empagliflozin / 750 mg Metformin XR FDC tablets: Experimental: low dose Empagliflozin/Metformin XR, 2 FDC tablets;
  1 x 25 mg tablet Empagliflozin / 3 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 3x Metformin XR tablets
- Total: Total of all reporting groups
Arm/Group | High Dose, Fasted | High Dose, Fed | Low Dose, Fasted | Total
Number analyzed (Participants) | 23 | 24 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (8.7) | 34.2 (9.2) | 30.8 (8.4) | 32.5 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 13 | 14 | 14 | 41

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration -Time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC 0-tz); Empagliflozin
Description: Area under the concentration -time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz); Empagliflozin
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1h 20min, 1h 40min, 2h, 2h 30min, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 16h, 24h, 36h, 48h and 72h after drug administration
Population: Pharmacokinetic set (PKS): This set includes all subjects of the Treated set (TS) who provided at least one observation for at least one primary endpoint and had no important protocol violations with respect to the statistical evaluation of Pharmacokinetic (PK) endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- High Dose, Fasted: 1 FDC Tablet: 1 FDC tablet, high dose, fasted: 25 mg Empagliflozin/1000 mg Metformin XR (extended release)
- High Dose, Fasted: 3 Single Tablets: 3 single tablets, high dose, fasted: 1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR
- High Dose, Fed: 1 FDC Tablet: 1 FDC tablet, high dose, fed: 25 mg Empagliflozin/1000 mg Metformin XR
- High Dose, Fed: 3 Single Tablets: 3 single tablets, high dose, fed: 1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR
- Low Dose, Fasted: 2 FDC Tablets: 2 FDC tablets, low dose, fasted: 12.5 mg Empagliflozin / 750 mg Metformin XR
- Low Dose, Fasted: 4 Single Tablets: 4 single tablets, low dose, fasted: 1 x 25 mg tablet Empagliflozin / 3 x 500 mg tablets Metformin XR
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24
nmol*h/L | 6430 (22.3) | 6430 (21.7) | 5690 (21.0) | 5850 (19.6) | 7160 (19.5) | 7110 (20.5)
Statistical Analysis 1: Comparison: High Dose, Fasted: 1 FDC Tablet vs High Dose, Fasted: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 99.98, 90% CI 2-sided [97.275 to 102.751], Standard Deviation 5.4 — Adjusted geometric mean (GM) ratio(%) was calculated as GM of 'High dose, fasted:1 FDC tablet' divided by GM of 'High dose, fasted:3 single tablets'.The 'standard deviation' is actually intra-individual geometric coefficient of variation (gCV (%))
Statistical Analysis 2: Comparison: High Dose, Fed: 1 FDC Tablet vs High Dose, Fed: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 97.09, 90% CI 2-sided [93.857 to 100.436], Standard Deviation 6.7 — The adjusted geometric mean ratio (%) was calculated as the geometric mean of 'High dose, fed: 1 FDC tablet' divided by the geometric mean of 'High dose, fed: 3 single tablets'. The 'standard deviation' is actually the intra-individual gCV (%)
Statistical Analysis 3: Comparison: Low Dose, Fasted: 2 FDC Tablets vs Low Dose, Fasted: 4 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 100.70, 90% CI 2-sided [98.28 to 103.18], Standard Deviation 4.9 — The adjusted geometric mean ratio (%) was calculated as the geometric mean of 'Low dose, fasted: 2 FDC tablets' divided by the geometric mean of 'Low dose, fasted: 4 single tablets'. The 'standard deviation' is actually the intra-individual gCV (%)

2. Primary Outcome: AUC 0-tz (Area Under the Concentration -Time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point); Metformin
Description: AUC 0-tz (area under the concentration -time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point); Metformin
Time Frame: as for outcome 1
Population: PKS: This set includes all subjects of the TS who provided at least one observation for at least one primary endpoint and had no important protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Low Dose, Fasted: 4 Single Tablets: 4 single tablets, low dose, fasted: 1 x 25 mg tablets Empagliflozin / 3 x 500 mg tablets Metformin XR
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Number analyzed (Participants) | 23 | 23 | 24 | 24 | 24 | 24
ng*h/mL | 6350 (32.8) | 6700 (28.9) | 13000 (23.6) | 13100 (21.1) | 10200 (38.5) | 10300 (38.3)
Statistical Analysis 1: Comparison: High Dose, Fasted: 1 FDC Tablet vs High Dose, Fasted: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0256, ANOVA; Adjusted geometric mean ratio (%) = 94.65, 90% CI 2-sided [82.29 to 108.88], Standard Deviation 28.1 — The adjusted geometric mean ratio (%) was calculated as the geometric mean of 'High dose, fasted: 1 FDC tablet' divided by the geometric mean of 'High dose, fasted: 3 single tablets'. The 'standard deviation' is actually the intra-individual gCV (%)
Statistical Analysis 2: Comparison: High Dose, Fed: 1 FDC Tablet vs High Dose, Fed: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 99.69, 90% CI 2-sided [96.25 to 103.26], Standard Deviation 7.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Low Dose, Fasted: 2 FDC Tablets vs Low Dose, Fasted: 4 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0020, ANOVA; Adjusted geometric mean ratio (%) = 99.76, 90% CI 2-sided [88.65 to 112.27], Standard Deviation 24.2 — [estimate comment as in outcome 1, analysis 3]

3. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity); Empagliflozin
Description: AUC 0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity); Empagliflozin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24
nmol*h/L | 6510 (22.9) | 6490 (21.6) | 5800 (21.8) | 5970 (20.5) | 7240 (19.7) | 7180 (20.8)
Statistical Analysis 1: Comparison: High Dose, Fasted: 1 FDC Tablet vs High Dose, Fasted: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 100.10, 90% CI 2-sided [97.555 to 102.719], Standard Deviation 5.1 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: High Dose, Fed: 1 FDC Tablet vs High Dose, Fed: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 97.01, 90% CI 2-sided [93.622 to 100.531], Standard Deviation 7.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Low Dose, Fasted: 2 FDC Tablets vs Low Dose, Fasted: 4 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 100.78, 90% CI 2-sided [98.36 to 103.27], Standard Deviation 4.9 — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma); Empagliflozin
Description: Cmax (maximum measured concentration of the analyte in plasma); Empagliflozin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24
nmol/L | 886 (27.3) | 810 (28.1) | 559 (29.0) | 601 (25.0) | 1010 (27.0) | 963 (29.7)
Statistical Analysis 1: Comparison: High Dose, Fasted: 1 FDC Tablet vs High Dose, Fasted: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0072, ANOVA; Adjusted geometric mean ratio (%) = 109.07, 90% CI 2-sided [99.892 to 119.100], Standard Deviation 17.4 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: High Dose, Fed: 1 FDC Tablet vs High Dose, Fed: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0004, ANOVA; Adjusted geometric mean ratio (%) = 92.42, 90% CI 2-sided [86.781 to 98.428], Standard Deviation 12.5 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Low Dose, Fasted: 2 FDC Tablets vs Low Dose, Fasted: 4 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0014, ANOVA; Adjusted geometric mean ratio (%) = 105.37, 90% CI 2-sided [96.600 to 114.942], Standard Deviation 17.7 — [estimate comment as in outcome 1, analysis 3]

5. Primary Outcome: Cmax (Maximum Measured Concentration of the Analyte in Plasma); Metformin
Description: Cmax (maximum measured concentration of the analyte in plasma); Metformin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Number analyzed (Participants) | 23 | 23 | 24 | 24 | 24 | 24
ng/mL | 822 (37.4) | 851 (28.8) | 1180 (27.4) | 1070 (22.8) | 1300 (34.4) | 1330 (41.3)
Statistical Analysis 1: Comparison: High Dose, Fasted: 1 FDC Tablet vs High Dose, Fasted: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0198, ANOVA; Adjusted geometric mean ratio (%) = 96.65, 90% CI 2-sided [83.337 to 112.079], Standard Deviation 29.8 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: High Dose, Fed: 1 FDC Tablet vs High Dose, Fed: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0007, ANOVA; Adjusted geometric mean ratio (%) = 110.17, 90% CI 2-sided [103.809 to 116.926], Standard Deviation 12.0 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Low Dose, Fasted: 2 FDC Tablets vs Low Dose, Fasted: 4 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0037, ANOVA; Adjusted geometric mean ratio (%) = 97.68, 90% CI 2-sided [86.942 to 109.734], Standard Deviation 23.8 — [estimate comment as in outcome 1, analysis 3]

6. Secondary Outcome: AUC 0-infinity (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity); Metformin
Description: AUC 0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity); Metformin
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Number analyzed (Participants) | 23 | 23 | 24 | 24 | 24 | 24
ng*h/mL | 6490 (35.2) | 6790 (29.6) | 13200 (24.0) | 13200 (21.6) | 10500 (41.9) | 10400 (39.9)
Statistical Analysis 1: Comparison: High Dose, Fasted: 1 FDC Tablet vs High Dose, Fasted: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0254, ANOVA; Adjusted geometric mean ratio (%) = 95.40, 90% CI 2-sided [82.42 to 110.44], Standard Deviation 29.4 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: High Dose, Fed: 1 FDC Tablet vs High Dose, Fed: 3 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p < 0.0001, ANOVA; Adjusted geometric mean ratio (%) = 99.63, 90% CI 2-sided [96.21 to 103.17], Standard Deviation 7.1 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Low Dose, Fasted: 2 FDC Tablets vs Low Dose, Fasted: 4 Single Tablets; Test type: Non-Inferiority or Equivalence — No formal testing; p = 0.0029, ANOVA; Adjusted geometric mean ratio (%) = 101.06, 90% CI 2-sided [89.70 to 113.86], Standard Deviation 24.4 — [estimate comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: From first trial medication intake until next intake or the end-of-trial visit, 10 days
Groups:
- High Dose, Fasted: 1 FDC Tablet: 1 fixed dose combination (FDC) tablet under fasted conditions:
  25 mg Empagliflozin/1000 mg Metformin XR (extended release), FDC: Experimental, high dose Empagliflozin/Metformin XR, FDC tablet
- High Dose, Fasted: 3 Single Tablets: 3 single tablets under fasted conditions:
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets
- High Dose, Fed: 1 FDC Tablet: 1 fixed dose combination (FDC) tablet under fed conditions:
  25 mg Empagliflozin/1000 mg Metformin XR, FDC: Experimental, high dose Empagliflozin/Metformin XR,FDC tablet
- High Dose, Fed: 3 Single Tablets: 3 single tablets under fed conditions:
  1 x 25 mg tablet Empagliflozin / 2 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 2x Metformin XR tablets
- Low Dose, Fasted: 2 FDC Tablets: 2 fixed dose combination (FDC) tablets under fasted conditions:
  12.5 mg Empagliflozin / 750 mg Metformin XR FDC tablets: Experimental: low dose Empagliflozin/Metformin XR, 2 FDC tablets
- Low Dose, Fasted: 4 Single Tablets: 4 single tablets under fed conditions:
  1 x 25 mg tablet Empagliflozin / 3 x 500 mg tablets Metformin XR: Active Comparator: 1x Empagliflozin / 3x Metformin XR tablets
Arm/Group | High Dose, Fasted: 1 FDC Tablet | High Dose, Fasted: 3 Single Tablets | High Dose, Fed: 1 FDC Tablet | High Dose, Fed: 3 Single Tablets | Low Dose, Fasted: 2 FDC Tablets | Low Dose, Fasted: 4 Single Tablets
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/23 | 1/23 | 1/24 | 2/24 | 4/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose, Fasted: 1 FDC Tablet (N=23) | High Dose, Fasted: 3 Single Tablets (N=23) | High Dose, Fed: 1 FDC Tablet (N=24) | High Dose, Fed: 3 Single Tablets (N=24) | Low Dose, Fasted: 2 FDC Tablets (N=24) | Low Dose, Fasted: 4 Single Tablets (N=24)
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.